CLINICAL TRIAL: NCT00637208
Title: Selective Retrograde Venography and Sclerotherapy of Internal Spermatic Veins and Associated Venous Bypasses and Retro-Peritoneal Collateral in Patients With Bilateral Varicocele and Localized Prostate Cancer
Brief Title: Sclerotherapy of Internal Spermatic Veins in Patients With Varicocele and Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maaynei Hayesha Medical Center (Other)
Responsible Party: Dr Uriel Levinger, Maaynei Hayesha Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVS-002-IL; MHMC grant
Record Dates: First submitted 2008-03-09; First posted 2008-03-17 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; venography; male patients; Localized microscopic prostate cancer up to Gleason 6 (3+3); PSA level <14; presence of varicocele
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: venographic occlusion of spermatic veins
- 2 (No Intervention): Watch-full follow-up

INTERVENTIONS:
Procedure: venographic occlusion of spermatic veins — Through the femoral vein a catheter is inserted into the spermatic veins in succession and the veins are occluded.
  Arms: 1

SUMMARY:
Patients with varicocele in whon early prostate cancer will be found will undergo venographic embolization of both spermatic veins. The study hypothesis is that this procedure will induce a gradual regression of the prostate volume that may decrease prostate cancer cells. Close follow-up will ensure that necessary therapy will be provided if needed according to clinical criteria. Results in terms of prostate size PSA level and tumor size will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Males age 45-75
* Prostate cancer
* Presence of varicocele
* No contraindication for venography

Exclusion Criteria:

* Diseases or medications which prevent interventional vascular procedures

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety performance of the procedure. The change in tumor size and prostate cancer cells as evaluated by trans-rectal ultrasound and prostate biopsy | one year

SECONDARY OUTCOMES:
The change in size of the prostate as evaluated by ultrasound Change in PSA value. Reduction of above 20% in nocturia | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Maaynei Hayesha Medical Center, Bnei Brak, Israel